CLINICAL TRIAL: NCT04330677
Title: Dissecting the Role of Estradiol in Mediating Gender-specific Anxiolytic and Prosocial Effects of Oxytocin
Acronym: ESMory
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Professor for Psychiatry, University of Oldenburg
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: ESMory
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Oxytocin; Estrogen; Fear Extinction; Emotion Processing; Memory
Keywords: fMRI; Oxytocin; Estrogen; Memory; Emotion Processing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. Oxytocin spray, 2. Estrogen gel (Experimental)
  Interventions: Drug: Oxytocin nasal spray; Drug: Estrogen Gel
- 1. Oxytocin spray, 2. Placebo gel (Experimental)
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo Gel
- 1. Placebo spray, 2. Estrogen gel (Experimental)
  Interventions: Drug: Placebo nasal spray; Drug: Estrogen Gel
- 1. Placebo spray, 2. Placebo gel (Placebo Comparator)
  Interventions: Drug: Placebo nasal spray; Drug: Placebo Gel

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal administration of 24 International Units, Oxytocin will be given 30 minutes before the fear extinction task (Study 1) or fMRI measurement (Study 2).
  Arms: 1. Oxytocin spray, 2. Estrogen gel; 1. Oxytocin spray, 2. Placebo gel
Drug: Placebo nasal spray — The placebo spray contains the identical ingredients, except for the peptide itself. It will be given 30 minutes before the fear extinction task (Study 1) or fMRI measurement (Study 2).
  Arms: 1. Placebo spray, 2. Estrogen gel; 1. Placebo spray, 2. Placebo gel
Drug: Estrogen Gel — Participants received a single dose of estradiol gel (Estramon 2 mg estradiol, Hexal AG, Holzkirchen, Germany), applied to their shoulder, 3 hours prior to the fear extinction task (Study 1) or fMRI measurement (Study 2).
  Arms: 1. Oxytocin spray, 2. Estrogen gel; 1. Placebo spray, 2. Estrogen gel
Drug: Placebo Gel — Participants received a single dose of the placebo gel (ultrasonic gel, 2 mg), applied to their shoulder, 3 hours prior to the fear extinction task (Study 1) or fMRI measurement (Study 2).
  Arms: 1. Oxytocin spray, 2. Placebo gel; 1. Placebo spray, 2. Placebo gel

SUMMARY:
The study aims to examine a behavioral and neural framework for understanding the sex-specific effects of the neuropeptide oxytocin (OXT). Using hormonal, behavioral and neuroimaging readouts, it is planned to explore the interplay of OXT and estradiol as a potential mechanism mediating sexual dimorphic effects.

DETAILED DESCRIPTION:
The study comprises two subprojects (Study 1 and Study 2). In Study 1, the investigators will compare the effects of OXT on fear extinction and fear recall as well as on emotion recognition between women and men. Additionally, the investigators plan to test whether a pretreatment with exogenous estradiol can be used to augment these OXT effects. In Study 2, the investigators will use functional magnetic resonance imaging (fMRI) to elucidate the effects of OXT-estradiol interactions on neural responses in an emotional face matching task and an emotional memory task. Half of the participants will be included in Study 1 and the other half in Study 2.

Study 1 contains three test sessions (after the screening). In the first session participants will complete a fear conditioning paradigm. The second session will take place on the following day and will start with the administration of estradiol gel (Divigel; 2 mg) or placebo (PLC). Three hours after the gel administration the participants will intranasally self-administer 24 IU of OXT or PLC under supervision and 30 min later a fear extinction task will commence, followed by an emotion recognition paradigm. A fear extinction recall task (identical with the fear conditioning task except for the electric shocks) will be conducted in the third session (with a 24-hours break between the second and the third session).

In Study 2, participants will be randomly assigned to four different treatment conditions (1. OXT + PLC gel; 2. OXT + estradiol gel; 3. PLC + PLC gel; 4. PLC + estradiol gel) after the screening session. The timing of the drug administration and blood sample collection will be identical to that of the second session of Study 1. The fMRI paradigms (resting state, emotional face matching and emotional memory) will start 30 minutes after nasal spray administration. Three days after the scanning, participants will be tested with a surprise recognition task, which includes pictures shown in the scanner and distractors.

ELIGIBILITY:
Inclusion Criteria:

* right handed
* healthy male & female volunteers
* women will be tested in their follicular phase (Day 0-5)

Exclusion Criteria:

* smoking
* pregnancy
* hormonal contraception
* current psychiatric illness
* current psychiatric medication or psychotherapy
* Study 2: MRI contraindication (e.g. metal in body, claustrophobia)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 487 (Actual)
Dates: Start 2016-09-18 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Electrodermal responses to fear-conditioned stimuli | 3 hours after gel administration and 30 minutes after nasal spray administration
  In Study 1, electrodermal responses will be measured during the fear conditioning and fear extinction tasks. The paradigm is an adapted version of a validated fear-conditioning procedure. Before the start of the paradigm a baseline of electrodermal activity is recorded for 60 seconds. During the conditioning session four neutral conditioned stimuli (two CS+ A and two CS+ B) are paired with an aversive US (electric shock) in 75 % contingency, whereas two other neutral stimuli are never paired with the US (non-fear-associated stimulus [CS-]). In CS+ trials electric shocks are administered during the last 500 milliseconds of the trial. In the fear extinction session all CS+ and CS- are presented in the absence of electric shocks. Oxytocin and estradiol baseline concentrations will be tested as moderator variables.
Emotion recognition thresholds | 200 minutes after gel administration and 50 minutes after nasal spray administration
  In Study 1, emotion recognition will be measured. During the emotion recognition task, emotional faces are presented and participants are required to indicate the perceived emotion ("neutral", "fearful", "happy", "disgusted", "angry", "not sure") in a following self-paced phase. A Bayesian adaptive procedure ("QUEST") will be used to determine the stimulus presentation and to estimate individual emotion thresholds. Oxytocin and estradiol baseline concentrations will be tested as moderator variables.
Resting state functional connectivity | 3 hours after gel administration and 30 minutes after nasal spray administration
  In Study 2, resting state functional connectivity will be measured. The resting state fMRI analysis will focus on functional connectivity between regions-of-interest (ROIs) associated with emotional processing (i.e. amygdala, cingulate and prefrontal cortex, insula, striatal areas). Oxytocin and estradiol baseline concentrations will be tested as moderator variables.
Neural responses to emotional faces | 190 minutes gel administration and 40 minutes after nasal spray administration
  In Study 2, neural responses to emotional faces will be measured. Functional magnetic resonance imaging will be performed to measure the blood-oxygen-level dependent signal in response to emotional faces. Analyses will focus on regions-of-interest associated with emotional processing (i.e. amygdala, cingulate and prefrontal cortex, insula, striatal areas). Oxytocin and estradiol baseline concentrations will be tested as moderator variables.
Neural responses to an emotional subsequent memory task | 200 minutes after gel administration and 50 minutes after nasal spray administration
  In Study 2, neural responses to an emotional subsequent memory task will be measured. Functional magnetic resonance imaging will be performed to measure the blood-oxygen-level dependent signal in response to emotional scenes. The investigators plan to analyze scenes depending on valence (positive, negative, neural) and sociality (social, non-social). Furthermore, remembered and non-remembered emotional pictures will be compared. To classify pictures as remembered and non-remembered, participants will perform a memory recognition task three days after the MRI scan. The recognition task will include pictures shown in the scanner and distractors. Analyses will focus on regions-of-interest associated with emotional processing and memory (i.e. amygdala, hippocampus, cingulate and prefrontal cortex, insula, striatal areas). Oxytocin and estradiol baseline concentrations will be tested as moderator variables.

SECONDARY OUTCOMES:
Changes in oxytocin plasma concentration | 5 minutes before gel administration and 5 minutes after the last task
  In both studies, blood samples will be collected 5 minutes before gel administration and 5 minutes after the last task.
Changes in estrogen plasma concentration | 5 minutes before gel administration and 5 minutes after the last task
  In both studies, blood samples will be collected 5 minutes before gel administration and 5 minutes after the last task.
Contingency ratings of fear-conditioned stimuli | 3 hours after gel administration and 30 minutes after nasal spray administration
  In Study 1, during the first 3500 ms of a trial in the fear conditioning and fear extinction tasks participants will be required to indicate via button press whether they expect to receive an electric shock (yes, no, not sure). Oxytocin and estradiol baseline concentrations will be tested as moderator variables.
Ultimatum game tasks | 150 minutes after gel administration
  In Study 1, bargaining behavior will be measured in three different versions of the Ultimatum Game (restricted, unrestricted and computer ultimatum game). All participants will play as responders in the three versions. As a cover story, participants will be told that they play against real partners, who took part in previous experiments. In the restricted version of the Ultimatum Game, the proposer can only decide between two given options. As such, chosen offers are either framed as fair or unfair depending on the alternative option. In the unrestricted Ultimatum Game, the proposer can freely decide how to split 10 Euro. In addition, participants will complete 24 trials of a computer version of the unrestricted Ultimatum Game, in which the word "computer" will be shown instead of a picture of the proposer. Estradiol baseline concentrations will be tested as moderator variables.
Delayed discounting task | 170 minutes after gel administration
  In Study 1, subjects will perform a delayed discounting task in order to assess their control of impulsive preferences. Participants will be asked to choose between small immediate rewards and larger later rewards. Estradiol baseline concentrations will be tested as moderator variables.
Changes in the Multifaceted Empathy Test (MET) | 135 minutes after the gel administration on the fMRI acquisition day and three days after the fMRI acquisition day
  In Study 2, participants' empathy will be assessed with the Multifaceted Empathy Test (MET) which includes photographs showing people in emotionally charged situations. Participants will be asked to infer the mental states of the individuals shown (cognitive empathy) and to rate their emotional response to the picture (emotional empathy). Participants will perform the MET twice: 1. before the fMRI in the second session and and 2. three days following the fMRI. Estradiol baseline concentrations will be tested as moderator variables.
Changes in the Prisoner's Dilemma | 155 minutes after the gel administration on the fMRI acquisition day and three days after the fMRI acquisition day
  In Study 2, the investigators will use an iterated version of the prisoner's dilemma to evaluate the participant's cooperative behavior. The participants will have to decide multiple times whether they want to betray their opponent or whether they choose to cooperate. Participants will perform the Prisoner's Dilemma twice: 1. before the fMRI in the second session and and 2. three days following the fMRI.Estradiol baseline concentrations will be tested as moderator variables.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Hurlemann, MSc, MD, PhD, Principal Investigator — University of Oldenburg
Locations (1):
- Deparment of Psychiatry and Medical Psychology, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hariri AR, Tessitore A, Mattay VS, Fera F, Weinberger DR. The amygdala response to emotional stimuli: a comparison of faces and scenes. Neuroimage. 2002 Sep;17(1):317-23. doi: 10.1006/nimg.2002.1179. PMID 12482086
- See also: Neuromodulation of Emotion (NEMO) research group — http://renehurlemann.squarespace.com/welcome/